CLINICAL TRIAL: NCT06447259
Title: A Rising Drug Burden Index, Not Anticholinergic Burden, is Related With Malnutrition in Community-dwelling Older Adults With Dementia
Brief Title: Drug Burden Index is Associated With Malnutrition in Community-dwelling Dementia Patients
Status: Completed | Type: Observational
Sponsor: Sultan Keskin Demircan (Other Government)
Responsible Party: Sponsor-Investigator, Sultan Keskin Demircan, Principal Investigator, Gulhane Training and Research Hospital
Organization: Gulhane Training and Research Hospital (Other Government)
Other Study IDs: GulhaneTR2
Record Dates: First submitted 2024-05-28; First posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2023-04

CONDITIONS: Malnutrition Severe; Dementia; Drug Use; Anticholinergic Toxicity
Keywords: Drug burden index,; older adults; malnutrition; anticholinergic drugs; dementia
MeSH Terms: conditions — Dementia; Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Malnutrition leads to poor clinical outcomes in dementia patients. The investigator aimed to examine the association between drug burden index (DBI) and anticholinergic burden (ACB) scores with nutrition status in community-dwelling older adults with dementia, considering that drugs may contribute malnutrition.

A total of 415 outpatients with dementia, evaluated by Mini Nutrition Assessment test and registered drug information, are included in the study. The investigator calculated the DBI as the sum of all sedatives and anticholinergics taken continuously for at least four weeks prior to admission and evaluated the ACB score.

Practice Impact: Due to accompanying chronic diseases and symptoms, cholinergic and/or sedative-loaded drugs are often prescribed to dementia patients. In this study, İnvestigators emphasized that in addition to the cholinergic loads of the drugs used, their sedative loads and the drug doses they use are also important. Avoiding prescribing these medications to patients with dementia will protect them from malnutrition and its negative consequences.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of any type of demantia
* Must be able to swallow tablets
* Must be recorded data of medications and doses

Exclusion Criteria:

* Psychiatric disorders
* Mild cognitive impairment
* End-stage diseases (renal, liver, cardiac)
* Uncontrolled thyroid functions

Ages: 65 Years to 100 Years | Sex: All
Age Groups: Older Adult
Study Population: The data of patients (65 years of age and older) who were applied to a tertiary geriatric outpatient clinic
Sampling Method: Non-Probability Sample
Enrollment: 415 (Actual)
Dates: Start 2023-05-20 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-12-10 (Actual)

PRIMARY OUTCOMES:
Number of participants with malnutrition, malnutrition risk and healthy | Baseline
  Based on the MNA-SF score, each participant was assigned to one of the following three groups: malnutrition (score between 0 and 7), malnutrition risk (score between 8 and 11), and healthy (score from 12 to 14).
Number of participants with high DBI (Drug Burden Index) score | Baseline
  Medications taken consistently at least four weeks prior to admission were considered to be in current use. DBI of drugs containing sedative and cholinergic load was calculated The following formula was used to calculate the DBI = D/ (δ +D), where D represents the daily dose consumed by participants and δ is the minimum recommended is the minimum daily dose that has been established in accordance with the adult dose authorized by the US Food and Drug Administration (FDA) and Turkish authorities in the product information of the drug. Each participant's total DBI score was determined by adding the DBI values for each substance with anticholinergic or sedative effects. Patients were classified as none (DBI=0), low exposure (0<DBI<1), or high exposure (DBI ≥1).
Number of participants with high ACB (Anti Cholinergic Burden) score | Baseline
  Medications taken consistently at least four weeks prior to admission were considered to be in current use.The anticholinergic drug exposure in each patient was assessed by a clinician using the Anticholinergic Cognitive Burden Scale, which grades the anticholinergic activity of each drug into three categories: absence (ACB = 0), possible (ACB = 1), and definite (either ACB = 2 or ACB = 3). The scores for each drug were added up to determine the patient's overall ACB score. All patients were then categorized into three groups: none (ACB score of 0), low to moderate exposure (ACB score of 1 or 2), or high exposure (ACB score of 3 or above)

CONTACTS AND LOCATIONS:
Locations (1):
- Sultan Keskin Demircan, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No